CLINICAL TRIAL: NCT05024656
Title: A Prospective, Multi-Center, Randomized Controlled, Parallel Group, Trial Evaluating the Use of AmnioExcel Plus Placental Allograft Membrane for the Management of Diabetic Foot Ulcers
Brief Title: AmnioExcel® Plus vs SOC in the Management of Diabetic Foot Ulcers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T-AEPDFU-002
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Diabetic Foot Ulcer
Keywords: diabetic foot; diabetes mellitus; diabetes complications
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Diabetes Complications | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, randomized, parallel-group Trial comparing the outcomes associated with the use of AmnioExcel® Plus Placental Allograft Membrane (AmnioExcel® Plus) used in conjunction with Standard of Care (SOC) compared to SOC alone in the management of diabetic foot ulcers (DFUs).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AmnioExcel Plus Amniotic Membrane + Standard of Care (Experimental): AmnioExcel Plus is a human placental-based tissue consisting of dehydrated, tri-layer Placental (Amnion/Chorion/Amnion) Allograft Membrane (T-PAM) layers. T-PAM is a minimally manipulated placental membrane product made from tissues donated by pre-screened mothers during planned C-sections and is intended for use as a wound covering in the homologous use for the repair, reconstruction and replacement of skin at the direction of a physician. AmnioExcel Plus contains Human Cellular and Tissue Based Products (HCT/P) as defined by US FDA 21 CFR Part 1271.
  Standard of care includes the following:
  * Coban™
  * Conforming gauze
  * Optifoam® non-adhesive dressing
  * Xtrasorb® for highly exudated wounds
  * Cotton Gauze
  * Normal saline (liquid or gel)
  * Non-adhering dressings
  * Steristrips
  * Offloading boot, as appropriate
  Interventions: Other: AmnioExcel Plus Amniotic Membrane; Other: Standard of Care
- Standard of Care (Active Comparator): * Coban™
  * Conforming gauze
  * Optifoam® non-adhesive dressing
  * Xtrasorb® for highly exudated wounds
  * Cotton Gauze
  * Normal saline (liquid or gel)
  * Steristrips
  * Offloading boot, as appropriate
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: AmnioExcel Plus Amniotic Membrane — AmnioExcel® Plus will be applied weekly, in conjunction with SOC, if the ulcer remains open, or up to and including Week 11, whichever comes first.
  Arms: AmnioExcel Plus Amniotic Membrane + Standard of Care
Other: Standard of Care — The dressings, materials, and appliances used in accordance with institutional protocol or professional clinical judgement.

SUMMARY:
This is a prospective, multicenter, randomized, parallel-group Trial comparing the outcomes associated with the use of AmnioExcel® Plus Placental Allograft Membrane (AmnioExcel® Plus) used in conjunction with Standard of Care (SOC) compared to SOC alone in the management of diabetic foot ulcers (DFUs).

DETAILED DESCRIPTION:
This study will have three (3) phases: (1) a Screening Phase, (2) a Treatment Phase, and (3) a Follow-up Phase. Subjects will be seen weekly in the Screening and Treatment Phases.

Subjects will be seen weekly in the Screening and Treatment Phases. Subjects who achieve confirmed wound closure during the Treatment Phase will be entered into the Follow-up Phase and will return to the site four (4) weeks following that confirmation visit.

ELIGIBILITY:
Inclusion Criteria:

* Have participated in the informed consent process and signed a study-specific informed consent document
* Be willing to comply with study procedures, including study visits, and compliance with study required off-loading/protective device for the duration of the study
* Be at least 18 years of age
* If female and of child-bearing potential, must not be pregnant. To document pregnancy status, subject statement is acceptable
* Have Type II or Type II diabetes mellitus with investigator-confirmed glycosylated hemoglobin (HbA1c) of less than or equal to 12% within 3 months prior to Screening Visit
* Have at least one diabetic foot ulcer that meets ALL the following criteria:

  1. Ulcer which has been in existence for a minimum of four weeks, prior to signing the Informed Consent Form allowing trial participation
  2. Ulcer is a partial or full thickness diabetic foot ulcer without capsule/tendon/bone exposure
  3. Ulcer does not have tunneling, undermining, or sinus tracts that necessitates surgical OR debridement and/or penetrates to capsule/tendon/bone
  4. Ulcer is located on the foot or ankle (with no portion above the top of the malleolus)
  5. Ulcer size (area) is greater than equal to 1 cm2 and less than equal to 12 cm2 post-debridement
* Have a minimum 4cm margin between the qualifying study ulcer and any other ulcer on that same foot, post-debridement

  (a) If the subject has more than one ulcer that meets eligibility criteria, the ulcer designated as the study ulcer will be at the discretion of the investigator
* Have adequate vascular perfusion of the affected limb as defined by at least one of the following within the past 60 days:

  1. Ankle-Brachial Index (ABI) greater than equal to 0.7 and less than equal to 1.2, performed within 60 days of screening,
  2. Toe pressure (plethysmography) > 40 mmHg at time of screening, or
  3. TcPO2 > 50 mmHg at time of screening
* Be willing and able to maintain required applicable dressing changes as well as study required off-loading/protective device for the duration of the study
* Have a study wound severity Wagner I or II

Exclusion Criteria:

* Previously randomized and treated under this clinical study protocol
* Patients with a known history of poor compliance with medical treatments
* Suspected or confirmed gangrene or ulcer infection of the study ulcer or is receiving systemic/IV antibiotics at the time of randomization
* Suspected or confirmed osteomyelitis of the foot with the study ulcer
* Participated in another clinical trial involving a device or a systemically administered investigational study drug/treatment within 28 days of randomization
* Received within 28 days of signing Informed Consent Form, or is scheduled to receive during study participation, a medication or treatment which is known to interfere with or affect the rate and quality of ulcer healing (e.g., systemic steroids, immunosuppressive therapy, autoimmune disease therapy, dialysis, radiation therapy to the foot, vascular surgery, angioplasty, or thrombolysis)
* History of bone cancer or metastatic disease of the affected limb, radiation therapy to the foot, or has had chemotherapy (i.e., systemic steroids, anti-rheumatics, TNF inhibitors, active chemotherapy, immunosuppressive therapy, autoimmune disease therapy) within 12 months prior to signing Informed Consent Form allowing trial participation
* In the opinion of the investigator, the subject has a history of, or is currently diagnosed with, any illness or condition, other than diabetes, that could interfere with ulcer healing (e.g., end-stage renal disease, severe malnutrition, liver disease, aplastic anemia, connective tissue disorder, acquired immune deficiency syndrome, HIV positive, or sickle cell anemia)
* In the opinion of the investigator, the subject has unstable Charcot foot or Charcot with bony prominence that could inhibit ulcer healing
* Have ulcers secondary to a disease other than diabetes (e.g., vasculitis, neoplasms, or hematological disorders)
* In the opinion of the investigator, the subject has excessive lymphedema that could interfere with off-loading and/or ulcer healing
* Study Ulcer has received ulcer dressings that included growth factors, engineered tissues, or skin substitutes within 28 days of randomization, or is scheduled to receive such treatment during the study (e.g., Regranex, Dermagraft, Apligraf, EpiFix, Grafix, GraftJacket, OASIS, Omnigraft, or Integra BMWD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of complete wound closure | Up to 12 weeks of treatment
  Number of wounds with complete wound closure as assessed by the investigator. Complete wound closure is defined as 100% re-epithelialization of the ulcer surface without detectable exudate.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Arnold, PhD, Study Director — Integra LifeSciences

IPD SHARING:
Plan to Share IPD: No